CLINICAL TRIAL: NCT00577772
Title: An Exploratory Assessment of Small Bowel Transit Time and Small Bowel Bacterial Overgrowth Using the SmartPill Capsule
Brief Title: Transit Time and Bacterial Overgrowth Using SmartPill Capsule
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment Goal Not Met
Sponsor: Mayo Clinic (Other)
Collaborators: The SmartPill Corporation (Industry)
Responsible Party: John DiBaise, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-002721
Record Dates: First submitted 2007-12-17; First posted 2007-12-20 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Small Bowel Bacterial Overgrowth; Gastrointestinal Diseases; Stomach Diseases; Digestive System Diseases
Keywords: SmartPill Capsule; Digestive System Diseases; Small Bowel Bacterial Overgrowth; Gastrointestinal Device; Oro-cecal
MeSH Terms: conditions — Gastrointestinal Diseases; Stomach Diseases; Digestive System Diseases | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Participants (Active Comparator): Healthy Participants will report for simultaneous lactulose hydrogen breath test (H_2BT) and SmartPill study after an overnight fast. They will swallow the SmartPill Capsule at the study site. After 4 hours, they will be allowed to leave the study site and consume their usual diet. They will return for removal of the data recorder 5 days later.
  Interventions: Device: SmartPill; Procedure: Lactulose hydrogen breath test (H_2BT)
- Symptomatic Participants (Active Comparator): Subjects with symptoms suggestive of small bowel bacterial overgrowth (SBBO) (e.g., diarrhea, bloating, abdominal discomfort) for at least 3 months will be divided into 2 groups based on the results of their previous testing for SBBO (5 SBBO positive patients, 5 SBBO negative patients).
  The symptomatic participants will report for simultaneous lactulose hydrogen breath test (H_2BT) and SmartPill study after an overnight fast. They will swallow the SmartPill Capsule at the study site. After 4 hours, they will be allowed to leave the study site and consume their usual diet. They will return for removal of the data recorder 5 days later.
  After the capsule has been demonstrated to be passed from the subject, the subjects with SBBO present will then enter into an open-label treatment using Rifaximin (400 mg PO TID) for 7 days.
  Interventions: Drug: Xifaxan; Device: SmartPill; Procedure: Lactulose hydrogen breath test (H_2BT)

INTERVENTIONS:
Drug: Xifaxan — Open-Label Treatment at 400 mg by mouth, 3 times a day, for 7 days; only for those symptomatic and positive SBBO patients.
  Other Names: Rifaximin
  Arms: Symptomatic Participants
Device: SmartPill — The SmartPill is a single-use, ingestible capsule that utilizes sensor technology to measure pressure, pH and temperature throughout the entire GI tract. The ACT-1 (SmartPill) GI Monitoring System includes an ingestible capsule, a receiver and video display software.
Procedure: Lactulose hydrogen breath test (H_2BT) — A hydrogen breath test provides information about the digestion of certain sugars or carbohydrates, such as milk sugar (lactose) or fruit sugar (fructose). The test is also used for detecting abnormal growth of bacteria within the small bowel by having the patient ingest lactulose.

SUMMARY:
The primary purpose of this exploratory study is to measure orocecal transit time using the SmartPill ambulant capsule technology and to compare this with the lactulose hydrogen breath test. Additionally, the ability of the SmartPill GI Monitoring System to discriminate between healthy human subjects and patients with small bowel bacterial overgrowth will be explored using analyses of both pH and pressure patterns within the stomach and small intestine. The study will be performed in both normal subjects and patients with and without small bowel bacterial overgrowth.

DETAILED DESCRIPTION:
Small bowel bacterial overgrowth (SBBO), an increasingly recognized malabsorptive condition caused by the excessive growth of bacteria in the small bowel, results in a spectrum of symptoms such as diarrhea, bloating abdominal discomfort and weight loss. Multiple factors both internal and external to the individual prevent excessive small bowel bacterial colonization and determine the types of bacteria present. The most important factors within the individual are normal small bowel motility, which prevents attachment of ingested organisms, and gastric acid, which destroys many organisms before they reach the small intestine. The determination of small bowel motility is problematic due to limitations of the tests available (e.g., hydrogen breath test, scintigraphy and manometry).

The SmartPill capsule is a recently developed novel device that, following its ingestion, can measure pH, pressure and temperature as it moves through the gastrointestinal tract. These recordings can be used to measure gastrointestinal transit and, potentially, other aspects of gastrointestinal motility/function. Previous studies using this device have demonstrated the ability of the SmartPill to measure the gastric residence time using the duration of acidic pH recording with good correlation between the gastric residence time of the SmartPill capsule and conventional gastric emptying scintigraphy.

ELIGIBILITY:
Inclusion Criteria for Healthy Subjects:

1. Mentally competent and able to give informed consent.
2. Healthy males and females between 18-70 years of age with no current or previous chronic gastrointestinal symptoms.

Inclusion Criteria for Symptomatic Subjects:

1. Males and females between 18-70 years of age with symptoms suggestive of small bowel bacterial overgrowth (e.g., diarrhea, bloating, abdominal discomfort) for at least 3 months during the previous 12 months (need not be consecutive) who recently underwent an evaluation for small bowel bacterial overgrowth by either hydrogen breath testing or culture of small bowel aspirate.
2. Ability to stop laxatives and prokinetic and narcotic analgesic agents 3 days prior to the study and during the study period.
3. Ability to stop proton pump inhibitors 7 days prior to the study and histamine type-2 receptor antagonists (H_2RAs) for 3 days prior to the study and during the study period.

Exclusion Criteria:

1. Subjects who are unable or unwilling to give informed consent or return for all required study visits.
2. Prior gastrointestinal surgery which has altered the anatomy of the esophagus, stomach or small/large intestine (exceptions include appendectomy, cholecystectomy and fundoplication).
3. Hypersensitivity to rifaximin.
4. Use of any medications in the previous week that could alter gastrointestinal motor function.
5. Body Mass Index (BMI) > 38.
6. Previous history of bezoars.
7. Any abdominal surgery within the past 3 months.
8. Known or history of inflammatory bowel disease.
9. History of diverticulitis, diverticular stricture, and other intestinal strictures.
10. Tobacco use within eight hours prior to capsule ingestion and during the initial 8 hour recording on the first day.
11. Alcohol use within eight hours prior to capsule ingestion and throughout the entire monitoring period (up to 5 days).
12. Females of childbearing age who are not practicing birth control and/or are pregnant or lactating (A urine pregnancy test will be performed on female subjects prior to capsule ingestion).
13. Cardiovascular, endocrine, renal or other chronic disease likely to affect motility.
14. Use of medical devices such as pacemakers, infusion pumps, or insulin pumps.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K. DiBaise, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: Healthy Participants will report for simultaneous lactulose hydrogen breath test (H_2BT) and SmartPill study after an overnight fast. They will swallow the SmartPill Capsule at the study site. After 4 hours, they will be allowed to leave the study site and consume their usual diet. They will return for removal of the SmartPill Capsule 5 days later.
- Symptomatic Participants: Subjects with symptoms suggestive of small bowel bacterial overgrowth (SBBO) (e.g., diarrhea, bloating, abdominal discomfort) for at least 3 months will be divided into 2 groups based on the results of their previous testing for SBBO (5 SBBO positive patients, 5 SBBO negative patients).
  The symptomatic participants will report for simultaneous lactulose hydrogen breath test (H_2BT) and SmartPill study after an overnight fast. They will swallow the SmartPill Capsule at the study site. After 4 hours, they will be allowed to leave the study site and consume their usual diet. They will return for removal of the SmartPill Capsule 5 days later.
  After the capsule has been demonstrated to be passed from the subject, the subjects with SBBO present will then enter into an open-label treatment using Rifaximin (400 mg PO TID) for 7 days.
Period: Overall Study
Arm/Group | Healthy Participants | Symptomatic Participants
Started | 10 | 7
Completed | 10 | 6
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Symptomatic Participants | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Oro-cecal Transit Time as Measured by SmartPill
Description: Oro-cecal transit time is the period of time needed by the head of the meal to reach the cecum, which is frequently used as an indicator of small intestinal transit time. Oro-cecal transit was to be determined simultaneously in the study subjects by both the SmartPill technique and the lactulose H_2BT technique.
Time Frame: baseline to passage of SmartPill, passage of SmartPill estimated no more than 72 hours from baseline
Population: Data were not analyzed as study was terminated early due to low enrollment.
Arm/Group | Healthy Participants | Symptomatic Participants
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each patient from baseline until the time that the SmartPill was eliminated from the body.
Arm/Group | Healthy Participants | Symptomatic Participants
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 6/10 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=10) | Symptomatic Participants (N=7)
Abdominal Pain/Cramping (Gastrointestinal disorders) | 2 (2) | 2 (2)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stress (Nervous system disorders) | 1 (1) | 0 (0)
Ankle Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intermittent vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper chest pain (General disorders) | 0 (0) | 1 (1)
Intermittent dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lodged SmartPill Capsule in Esophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early because enrollment goals were not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes